CLINICAL TRIAL: NCT05921396
Title: Assessment of Nasal Obstruction, a Comparison Between Rhinomanometry and Nasal Inspiratory Peak Flow at Patients After Endoscopic Nasal Surgery
Brief Title: Nasal Obstruction Compared by Rhinomanometry and Nasal Inspiratory Peak Flow After Endoscopic Nasal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Collaborators: University of Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FNO/2023/RMM-NPIF
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Pituitary Adenoma Invasive; Nasal Obstruction
Keywords: Pituitary Adenoma; Nasal surgery; Rhinomanometry; Nasal inspiratory peak flow; Endoscopic nasal surgery
MeSH Terms: conditions — Nasal Obstruction; Pituitary Neoplasms

STUDY DESIGN:
Intervention Model Description: The study subjects will be enrolled into one study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nasal patency before and after pituitary adenoma surgery (Experimental): Nasal patency in patients with pituitary adenoma indicated to endoscopic transnasal extirpation of the pituitary adenoma.
  Interventions: Procedure: Nasal patency - rhinomanometry; Procedure: Nasal patency - nasal inspiratory peak flow

INTERVENTIONS:
Procedure: Nasal patency - rhinomanometry — Nasal patency before and after the pituitary adenoma surgery will be assessed using rhinomanometry.
Procedure: Nasal patency - nasal inspiratory peak flow — Nasal patency before and after the pituitary adenoma surgery will be assessed using nasal inspiratory peak flow..

SUMMARY:
The aim of the project is to determine whether nasal inspiratory peak flow is sufficient for preoperative and postoperative measurement of nasal patency compared to rhinomanometry.

DETAILED DESCRIPTION:
The nasal cavity is used to heat, humidify and purify the air before entering other parts of the respiratory system. Other functions of the nose include in particular olfactory, immune, reflex, or sexual functions. Proper airflow through the nasal cavity is essential for all nasal functions; anatomical or flow changes can significantly affect nasal functions.

Endoscopic transnasal surgical approaches are modern, mini-invasive methods, enabling the solution of pathologies in the area of the cranial base, through the nasal cavity. The advantage of this technique is the absence of external incisions and scars and significantly better cosmetic effect, these methods also offer very good clarity and illumination of the operating field. The main disadvantage is the risk of affecting the functions of the nose. To create a transnasal approach to the skull base, it is necessary to perform lateralization of middle turbinates, resection of the anterior wall of the sphenoidal sinus, and resection of the posterior part of the nasal septum. These interventions are necessary for a good overview and manipulation in the operated area, however, they can lead to postoperative changes in the physiological functions of the nasal cavity, especially loss of smell, and taste, altered airflow through the nasal cavity, mucociliary transport disorders, nasal obstruction, crusting or drying mucous membrane. All these adverse changes significantly affect the patient's quality of life.

As a standard, rhinomanometry is used to measure nasal patency before and after surgery. A modern new method is measuring the patency of the nasal cavity using an NPIF (nasal peak inspiratory flow) device, which has significantly lower acquisition costs, is easy to use, and, above all, fast. The disadvantage is that the examination is less detailed, the result is the amount of air flowing in l/min through the nasal cavity.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* patients with pituitary adenoma indicated to endoscopic transnasal extirpation of the pituitary adenoma

Exclusion Criteria:

* patients after surgery of the nasal cavity or base of the skull
* patients with nasal disease and paranasal sinuses
* patients with olfactory disorders before surgery
* patients with nasal septal deviation that requires septoplasty

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of nasal patency measurement using rhinomanometry and NPIF | 3 months
  Comparison of nasal patency measurement using rhinomanometry and Nasal Peak Inspiratory Flow (NPIF) will be performed at the preoperative examination, 1 month and 3 months after surgery. The volume will be measured in L/min.
  Rhinomanometry is a standard diagnostic tool aiming to objectively evaluate the respiratory function of the nose. It measures pressure and flow during normal inspiration and expiration through the nose.
  Nasal peak inspiratory flow (NPIF) measures the maximum airflow a patient is able to produce during forced nasal inspiration and is a measure of nasal patency.

SECONDARY OUTCOMES:
Olfactory examination | 3 months
  Olfactory examination (test of identification and discrimination with perfumed markers) will be performed at the preoperative examination, 1 month and 3 months after surgery.
Lund-Kennedy scoring system | 3 months
  Evaluation of the nasal cavity and patency using the Lund-Kennedy scoring system (evaluation of edema, secretion, crust) will be performed at the preoperative examination, 1 month and 3 months after surgery. The total scores will be compared. The Lund-Kennedy score is a validated scale by which physicians rate the endoscopic appearance of the sinonasal cavity. There are 5 parameters rated on a scale of 0-2 for each side of the nose, for a maximum total score of 20 points. A higher score represents a worse endoscopic appearance.
SNOT 22 questionnaire | 3 months
  Sino-Nasal Outcome Test-22 (SNOT 22) Questionnaire (version 4) - patients will complete a list of symptoms and social/emotional consequences of their nasal disorder. The SNOT-22 is a validated scale that measures sinonasal symptoms in patients with sinusitis. The 22 questions are scored on a scale of 0-5 with a maximum total score of 110. Higher scores represent more symptomatic patients.
RhinoVAS questionnaire | 3 months
  Rhino Visual Analogue Scale (RhinoVAS) questionnaire will be used to assess postoperative changes in nasal function ranging from 0 (complete nose patency) to 10 cm (complete nose obstruction).
Nose Score | 3 months
  A simple, five-question, validated survey that uses a 20-point scale to capture breathing symptoms, with higher scores indicating more severe symptoms than lower scores. A score of 0 means no problems with nasal obstruction and a score of 100 means the worst possible problems with nasal obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Lubojacký, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Messerer M, Cossu G, George M, Daniel RT. Endoscopic Endonasal Trans-sphenoidal Approach: Minimally Invasive Surgery for Pituitary Adenomas. J Vis Exp. 2018 Jan 17;(131):55896. doi: 10.3791/55896. PMID 29364265
- [Background] Regmi D, Thapa A, Kc B, Shakya B. Endoscopic Endonasal Transsphenoidal Approach to Pituitary Adenoma: A Multi-disciplinary Approach. J Nepal Health Res Counc. 2017 Sep 8;15(2):174-177. doi: 10.3126/jnhrc.v15i2.18209. PMID 29016590
- [Background] Rochet M, El-Hage W, Richa S, Kazour F, Atanasova B. Depression, Olfaction, and Quality of Life: A Mutual Relationship. Brain Sci. 2018 May 4;8(5):80. doi: 10.3390/brainsci8050080. PMID 29734670
- [Background] Croy I, Nordin S, Hummel T. Olfactory disorders and quality of life--an updated review. Chem Senses. 2014 Mar;39(3):185-94. doi: 10.1093/chemse/bjt072. Epub 2014 Jan 15. PMID 24429163
- [Background] Schreiber A, Bertazzoni G, Ferrari M, Rampinelli V, Verri P, Mattavelli D, Fontanella M, Nicolai P, Doglietto F. Nasal Morbidity and Quality of Life After Endoscopic Transsphenoidal Surgery: A Single-Center Prospective Study. World Neurosurg. 2019 Mar;123:e557-e565. doi: 10.1016/j.wneu.2018.11.212. Epub 2018 Dec 5. PMID 30528530
- [Background] Rotenberg B, Tam S, Ryu WH, Duggal N. Microscopic versus endoscopic pituitary surgery: a systematic review. Laryngoscope. 2010 Jul;120(7):1292-7. doi: 10.1002/lary.20949. PMID 20578228
- [Background] Soyka MB, Serra C, Regli L, Meier E, Holzmann D. Long-term olfactory outcome after nasoseptal flap reconstructions in midline skull base surgery. Am J Rhinol Allergy. 2017 Sep 1;31(5):334-337. doi: 10.2500/ajra.2017.31.4463. PMID 28859712